CLINICAL TRIAL: NCT02853617
Title: A Phase I/II, Single and Repeat Dose, Dose Escalation Study of AV0328 Administered to Healthy Adult Volunteers
Brief Title: A Study of AV0328 Administered to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alopexx Vaccine, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AV-101-16
Record Dates: First submitted 2016-07-21; First posted 2016-08-03 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: PNAG-expressing Pathogenic Microbes Vaccine
Keywords: S. pneumoniae; N. meningitidis; H. influenza; B. pertussis; C. tetani; MRSA
MeSH Terms: conditions — Tetanus | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- AV0328 - Cohort 1 (Experimental): Cohort 1 will receive 15 µg to be given as an IM injection
  Interventions: Biological: AV0328 - Cohort 1
- AV0328 - Cohort 2 (Experimental): Cohorts 2 will receive 30 µg to be given as an IM injection
  Interventions: Biological: AV0328 - Cohort 2
- AV0328 - Cohort 3 (Experimental): Cohorts 3 will receive 75 µg to be given as an IM injection
  Interventions: Biological: AV0328 - Cohort 3
- AV0328 - Cohort 4 (Experimental): Cohorts 4 will receive 150 µg to be given as an IM injection
  Interventions: Biological: AV0328 - Cohort 4

INTERVENTIONS:
Biological: AV0328 - Cohort 1 — Cohort 1 will receive 15 µg to be given as an IM injection
  Other Names: study drug
  Arms: AV0328 - Cohort 1
Biological: AV0328 - Cohort 2 — Cohort 2 will receive 30 µg to be given as an IM injection
  Other Names: study drug
  Arms: AV0328 - Cohort 2
Biological: AV0328 - Cohort 3 — Cohort 3 will receive 75 µg to be given as an IM injection
  Other Names: study drug
  Arms: AV0328 - Cohort 3
Biological: AV0328 - Cohort 4 — Cohort 4 will receive 150 µg to be given as an IM injection
  Other Names: study drug
  Arms: AV0328 - Cohort 4

SUMMARY:
AV0328 is a novel vaccine candidate intended to raise antibodies to the glucosamine backbone of naturally occurring Poly N-acetyl glucosamine (PNAG), a capsular polysaccharide expressed on the surface of a wide array of microbes.

AV-101-16: A single and repeat dose, dose-escalation phase I/II study to evaluate the safety of intramuscularly administered AV0328. Approximately 16 subjects will be enrolled at a single U.S. center, based on 4 subjects per dose group. The study will consist of 3 parts: Part 1 will be a single dose, dose escalation study; Part 2 will assess the effect of a second dose of AV0328; Part 3 will assess the ability of a booster injection of AV0328 at Month 6 to restore protective titers against N. meningitidis B16B6 bacteria.

DETAILED DESCRIPTION:
AV0328 is a novel vaccine candidate intended to raise antibodies to the glucosamine backbone of naturally occurring Poly N-acetyl glucosamine (PNAG), a capsular polysaccharide expressed on the surface of a wide array of microbes.

AV-101-16: A single and repeat dose, dose-escalation phase I/II study to evaluate the safety of intramuscularly administered AV0328. Approximately 16 subjects will be enrolled at a single U.S. center, based on 4 subjects per dose group. The study will consist of 3 parts: Part 1 will be a single dose, dose escalation study; Part 2 will assess the effect of a second dose of AV0328; Part 3 will assess the ability of a booster injection of AV0328 at Month 6 to restore protective titers against N. meningitidis B16B6 bacteria.

Part 1 - Single Administration of AV0328:

Following injection, subjects will be observed for 28 days to determine the safety and tolerability of a single administration of AV0328. Cohort 1 will receive 15 µg to be given as an IM injection on Day 1. Cohorts 2, 3 and 4 will receive 30, 75 and 150 µg, respectively. The first subject of each cohort must be observed for a minimum of 24 hours before the remaining subjects in that group can be treated.

Dosage escalation will occur only after the final subject at each dose level has been observed for a minimum of 2 days and no dose limiting drug-related toxicity has occurred.

Part 2 - Second Administration of AV0328:

Following review of safety and tolerance for a minimum of 22 days of Part 1 by the Safety Review Committee (SRC), subjects from each dose level will return to receive an additional injection at the same dose level of AV0328 on Day 29. Additional safety and pharmacodynamic (PD) data will be collected through Week 52.

Part 3 - Booster Administration of AV0328 Serum drawn at Day 57 revealed that 3 of 4 subjects in Cohort 3 and all 4 subjects in Cohort 4 achieved protective titers against N. meningitidis B16B6 bacteria, defined as >30% killing at a titer of 1:8 or greater by BSA. If those titers fall below protective levels in a subject at 4 or 6 months, that subject will receive a booster injection at the 6-month time point or shortly thereafter. The dose will be 150 µg, IM which will be formulated in the same manner as the 150 µg dose in Parts 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteer.
2. Age 18-55 years, inclusive.
3. Normal hematological, hepatic, and renal function.
4. Subjects participating in the study are to use adequate birth control measures (abstinence, oral contraceptives, barrier method with spermicide or surgical sterilization) during study participation. Females of childbearing potential must have a negative pregnancy test on the days of dosing. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months.
5. If subject is female and of childbearing potential, she has a negative serum pregnancy test during screening and baseline and must be willing to undergo urine pregnancy testing during the study.
6. Subject must sign written informed consent and be willing and able to comply with protocol requirements.
7. Subject must be accessible for repeat dosing and follow-up.

Exclusion Criteria:

1. Major organ dysfunction.
2. Any significant pre-existing condition preventing full compliance with the study.
3. Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization for worsening disease within 3 months before receipt of study vaccine.
4. Allergic to vaccine components of AV0328, including poly N-acetyl glucosamine (PNAG), tetanus toxoid (TT) or alum; any previous severe reaction to any TT vaccine including arthus-type hypersensitivity reaction.
5. Vaccinations within one month prior to participation or 2 months after enrollment.
6. Women who are pregnant or lactating.
7. Abnormal skin or tattoo overlying the deltoid muscle in the immediate vicinity of the anticipated injection sites.
8. Donation of blood volume of 250 mL or greater or donation of plasma within 3 months prior to enrollment through conclusion of the study.
9. Bleeding condition associated with prolonged bleeding time that may contraindicate intramuscular (IM) injection or blood draw including subjects taking anticoagulant, antiplatelet and/or antithrombotic agents except for low-dose daily aspirin within 30 days before enrollment through completion Day 57.
10. Subjects currently on immunosuppressive or immunomodifying therapy or with a history of immunosuppressive or immunomodifying therapy (including systemic glucocorticoid therapy within 30 days of .AV0328 administration) .
11. Participation in other investigational or interventional studies within 30 days before the current study begins and/or during study participation. Participation in purely observational studies is acceptable.
12. Known active disease with human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV), or positive screening test for HIV, HBV and/or HCV.
13. A prior history of brachial neuritis, Guillan-Barre syndrome or other serious neurologic illness.
14. Prior severe staphylococcal infection or bacteremia.
15. Any clinically significant abnormality in any screening or Baseline laboratory test or electrocardiogram (ECG).
16. Medical condition or circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol or the subject's well-being or safety.

In addition, any patient who has met all of the eligibility criteria and has been enrolled in the study who subsequently experiences an acute febrile illness, must be afebrile for at least two days before administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events (AEs) at Day 57 following AV0328 vaccination | Day 1 through Day 57
  Continuous safety and tolerability monitoring of escalating doses of AV0328 in healthy adult volunteers at Day 57 with special attention to changes in bowel habits

SECONDARY OUTCOMES:
Serologic evidence of efficacy of AV0328 against S. pneumoniae, N. meningitidis, and methicillin-resistant S. aureus at Day 57 | Pre-dose, Days 29 and 57
  Serologic evidence of efficacy measured by pharmacodynamic blood biomarkers

OTHER OUTCOMES:
Serologic evidence of efficacy against other PNAG-expressing pathogens | Day 1 through Day 57
  Serologic evidence of efficacy measured by pharmacodynamic blood biomarkers
Number of patients with adverse events, including any newly diagnosed chronic conditions, up to Month 18 | Day 1 through Month 18
  Additional safety monitoring of escalating doses of AV0328 in healthy adult volunteers up to Month 18
Serologic evidence of efficacy up to Month 18 | Day 1 up to Month 18
  Additional serologic evidence of efficacy measured by pharmacodynamic blood biomarkers up to Month 18
Restore serologic protection against N. meningitidis B16B6 | Month 12
  Serologic evidence of efficacy measured by pharmacodynamic blood biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Hal Landy, MD, Study Director — Alopexx Vaccine, LLC
Locations (1):
- Inflamax Research, Inc., Neptune City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No